CLINICAL TRIAL: NCT02265263
Title: Biomarker Development for Postoperative Cognitive Impairment in the Elderly (BioCog)
Acronym: BioCog
Status: Terminated | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Claudia Spies, Univ.-Prof. Dr. med. C. Spies, Charite University, Berlin, Germany
Other Study IDs: BioCog
Record Dates: First submitted 2014-09-23; First posted 2014-10-15 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Delirium (POD); Postoperative Cognitive Deficit (POCD)
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Whole blood-/plasma (RNA-/DNA-Analysis)
  * Cerebrospinal fluid (sequencing of candidate nicotinic receptor genes and genes for acetylcholine synthesis/-catabolism: CHRNA3, CHRNA4, CHRNA5, CHRNA7, CHRNB2, CHRNB4, ACHE, CHAT) (only in Berlin).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Surgical patients - 3 Tesla MRI: A study group of at maximum n= 1200 is collected for measuring 3 Tesla MRI at two timepoints (Baseline and 90 days) in Berlin/Utrecht. They include surgical procedures within body cavity e.g. abdomen or thorax from departments of general surgery, urology, gynecology or thoracic surgery; orthopaedic operations (hip-, knee-, endoprosthesis or spine (including neurosurgical spine operations)); cardiac surgery and operation of extracranial/intracranial head and neck
  Data collection from study center Utrecht ist within one year after initial hospital stay. Data collection from study center Berlin is within two years after initial hospital stay.
- Patients ASA II/III - 3 Tesla MRI: A control group of at maximum n= 300 ASA II/III- patients is collected for measuring the learning experience during the cognitive testings. They are matched on age, education, and gender to the study patients. The 104 ASA II/III- patients should receive additionally MRI-scan (3 Tesla) at baseline, after 3 months and after 1 year in Utrecht, after 3 months, after 1, 2 years in Berlin.
  Data collection from study center Utrecht ist within one year after initial hospital stay. Data collection from study center Berlin is within five years after initial hospital stay.
- Volunteers ASA I/II - 3 Tesla MRI: To analyze scanner variability we additionally measure at maximum 20 subjects (Age ≥ 65 years) from Utrecht in the MRI scanner (3-Tesla) in Berlin and vice versa.
- Surgical patients - 7 Tesla MRI: A study Group of at maximum n= 80 should be collected for measuring 7 Tesla MRI at two timepoints (Baseline and 90 days) in Berlin.

SUMMARY:
The research leading consortium to these results has received funding from the European Union Seventh Framework Programme [FP7/2007-2013] under grant agreement no 602461 (www.biocog.eu).

The investigators will establish valid biomarkers panels (neuroimaging and molecular) for risk and clinical outcome prediction of postoperative delirium (POD)/postoperative cognitive deficit (POCD) in elective surgical patients (Age ≥ 65 years) in study centers in Berlin,Germany (data collection within 2 years after initial hospital stay) and Utrecht, The Netherlands (data collection within 1 year after initial hospital stay), thereof cerebrospinal fluid (only once on day of surgery in patients with planned spinal anesthesia/combined spinal epidural analgesia in patients, only in Berlin).

A control group of ASA II/III- patients is collected for measuring the learning experience during the cognitive testings. The participants are matched on age, education, and gender to the study patients. The ASA II/III- control patients receive additionally MRI-scan (3 Tesla) at baseline, after 3 months and after 1 (Utrecht) and 2 years (Berlin).

To analyze scanner variability we additionally measure at maximum 20 subjects (Age ≥ 65 years, ASA I and II) from Utrecht in the MRI scanner (3-Tesla) in Berlin and vice versa.

A study group at maximum (n= 80) and is collected for measuring 7 Tesla MRI at two timepoints (Baseline and 90 days).The primary endponit of this substudy is gamma amino-butyric acid concentration in CNS after 3-months (measured by MRI). A retrospective comparison group (extracting 8000 intensive care unit patient data from the patient data management system during the BioCog study period in 2016) to analyse economic effects that are caused by the implementation of quality indicators in health care.

An interim-analysis is performed on the primary endpoint after 400 included patients.

The resulting (multivariate) expert system is expected: 1) to support clinical decision-making in patient care, e.g. to balance the individual POD/POCD risk against the expected overall clinical outcome of an (elective) surgical intervention, 2) to allow the design of more sophisticated and hypothesis-driven clinical studies and drug trials (translational research) in the future. The latter will be possible on the basis of biomarker-based sub-grouping of patients and a better understanding of relevant pathophysiological processes.

Furthermore, a state-of-the art clinical database and biobank will be created that does not yet exist worldwide. Both the expert system and the reference database/biobank will expand the leadership of the contributing academic institutions in this particular research area. In addition, the newly created biobank will become an integral part of the European Biobanking and Biomolecular Resources Research Infrastructure (BBMRI) which allows top address specific and hypothesis-driven research questions.

Most notably, the developed (multivariate) expert system also has the potential for commercialization. Possible customers are: 1) physicians and hospital departments being involved in pre-surgical decision making, 2) pharmaceutical industry intending to conduct biomarker-based drug trials in POD/POCD.

ELIGIBILITY:
Study Group (Berlin/Utrecht):

Inclusion Criteria:

* Male and female patients aged ≥ 65 years, of European descent (Caucasian)
* Elective surgery with an expected operative time ≥ 60 minutes
* Ability to give informed consent after receiving spoken and written information of the study
* Eligibility for magnetic resonance Imaging

Exclusion Criteria:

* Mini-Mental-State-Examination ≤ 23 points
* Homelessness or other circumstances where the patient would not be reachable by phone or postal services during follow-up.
* Participation in another prospective interventional clinical study during participation in this clinical study during hospital stay
* Accommodation in an institution due to an official or judicial order
* Missing informed consent for saving and hand out pseudonymous data
* Neuropsychiatric morbidity, which limits the conduction of the neurocognitive testing
* Anacusis or Hypoacusis, which limits the conduction of the neurocognitive testing

Intraoperative clectroencephalography - examinations (Study Group Berlin):

Exclusion criteria:

* Neurological preconditions
* Proposed neurological surgery

Control Group (Berlin/Utrecht):

Inclusion criteria:

* Male and female patients aged ≥ 65 years, of European descent (Caucasian)
* ASA II and III patients
* No operation in the last half year before study inclusion
* Eligibility for magnetic resonance Imaging

Exclusion Criteria:

* Mini-Mental-State-Examination ≤ 23 Points
* Missing informed consent for saving and hand out pseudonymous data
* Neuropsychiatric morbidity, which limits the conduction of the neurocognitive testing
* Anacusis or Hypoacusis, which limits the conduction of the neurocognitive testing
* Taking psychothropic drugs (including sleep-inducing drug and benzodiazepine) on a regular basis and substances, which limit the conduction of the neurocognitive testing

Control Group (Utrecht) - Scannervariability:

Inclusion criteria:

* Male and female patients aged ≥ 65 years, of European descent (Caucasian)
* ASA I and II patients
* No operation in the last half year before study inclusion
* Eligibility for magnetic resonance Imaging

Study Group (Berlin) - 7 Tesla MRI:

Criteria as of the 3-Tesla- study group and additionally:

Exclusion criteria:

* absolute 7 - Tesla MRI-contraindications
* relative 7 - Tesla MRI-contraindications

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Surgical patients, 65 years or above (Berlin/Utrecht) ASA I and II patients, 65 years or above (Utrecht) ASA II and III patients, 65 years or above (Berlin/Utrecht)
Sampling Method: Non-Probability Sample
Enrollment: 1054 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium | Participants will be followed for the duration of hospital stay, an expected average of 7 days
  Postoperative delirium rate, defined according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) and/or as ≥ 2 cumulative points in the nursing Delirium Screening Scale (Nu-DESC) and/or a positive Confusion Assessment Method (CAM) and/or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) score and/or patient chart review that shows descriptions of delirium.
Incidence of postoperative cognitive deficit (POCD) | Up to 3 months after the operation
  POCD will be measured by a defined Cambridge Neuropsychological Test Automated Battery (CANTAB) POCD will be measured by a defined Cambridge Neuropsychological Test Automated Battery (CANTAB) and paper pencil tests (TMT A und B, Grooved Pegboard) and the Mini - Mental State Examination (MMSE)

SECONDARY OUTCOMES:
Duration of Delirium | Participants will be followed for the duration of hospital stay, an exspected average of 7 days
  * Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
  * Nursing Delirium Screening Scale (Nu-DESC)
  * Intensive Care Delirium Screening Checklist (ICDSC)
  * Delirium Detection Scale (DDS)
  * Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)
  * Confusion Assessment Method (CAM)
  * Chart Review
Duration of subsyndromal postoperative delirium | Participants will be followed for the duration of hospital stay, an exspected average of 7 days
  Nu-DESC score 1 and/or any criteria suggestive of POD (as described under "Primary Outcome Measures") that do not fulfill DSM-5 criteria for delirium.
Incidence of subsyndromal postoperative delirium | Participants will be followed for the duration of hospital stay, an exspected average of 7 days
  Nu-DESC score 1 and/or any criteria suggestive of POD (as described under "Primary Outcome Measures") that do not fulfill DSM-5 criteria for Delirium
Intensive care unit length of stay | Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
Hospital length of stay | Participants will be followed for the duration of hospital stay, an exspected average of 7 days
Postoperative organ complications | Participants will be followed for the duration of hospital stay, an exspected average of 7 days
  Postoperative organ complications are classified according to Clavien - Dindo classification.
Incidence of postoperative cognitive deficit | 1 year, 2 years, 5 years after the operation
  POCD will be measured by a defined Cambridge Neuropsychological Test Automated Battery (CANTAB), paper pencil tests (TMT A und B, Grooved Pegboard) and the Mini - Mental State Examination (MMSE)
Socioeconomic characteristics | 3 months, 1, 2 and 5 years after the operation
  Study center Berlin: Health economic data according to cost of patient care (The §21 dataset (diagnoses and operation-codes). Hospital costs are calculated according to the Institute for the Hospital Remuneration System (InEK) calculation scheme to compare the refinanced costs in each cost category/cost-center segment from study center Charité. Necessity and indirect costs of medical care (outpatient visits) after hospital stay.
Health related quality of life | 3 months, 1, 2 and 5 years after the operation
  Study center Berlin: Measurement by EQ-5D
Barthel Index | 3 months, 1, 2 and 5 years after the operation
Instrumental activities of daily living scale | 3 months, 1, 2 and 5 years after the operation
Hand grip strength test | 3 months, 1, 2 and 5 years after the operation
Malnutrition | 3 months, 1, 2 and 5 years after the operation
  Mini Nutritional Assessment - Short form, Serum albumin
Mobility | 3 months, 1, 2 and 5 years after the operation
  Timed up and go test
Neuroimaging Biomarker | 3 months, 1, 2 and 5 years after the operation
Molecular Biomarker | 3 months
Health related Quality of life | 3 months, 1 year after the operation
  Study center Utrecht: Measurement by EQ-5D
Socioeconomic characteristics | 3 months, 1 year after the operation
  Study center Utrecht: Health economic data according to direct cost of patient care (inpatient and outpatient stays) and necessity and indirect costs of medical care (outpatient visits) after hospital stay.
Heart rate variability | Study center Berlin: Participants will be followed for the duration of hospital stay, an exspected average of 7 days
Light Levels (lux) | Study center Berlin: Participants will be followed for the duration of hospital stay, an exspected average of 7 days
Light frequencies | Study center Berlin: Participants will be followed for the duration of hospital stay, an exspected average of 7 days
Depression | Participants will be followed for the duration of hospital stay, an exspected average of 7 days
  Hospital Anxiety and Depression Scale (HADS) (Study Center Utrecht), GDS-15 (Study Center Berlin)
Anxiety | Participants will be followed for the duration of hospital stay, an exspected average of 7 days
  Faces Anxiety Scale (FAS)
Electroencephalography (EEG)- Mapping | At time of surgery
  Study center Berlin: EEG with19 electrodes and hypo- and hyperventilation in physiological limits (no patients with neurological pre-existing conditions or proposed neuro-surgery)
Mortality | 3 months, 1, 2 and 5 years after the operation
Depth of consciousness index | At time of surgery
  Depth of consciousness index measured by processive Electroencephalography and Electromyography (EEG/EMG) -Data (SedLine®)
Intraoperative cerebral oxymetry | At time of surgery
Changes of Electroencephalography | Participants will be followed up until the end of postanesthesia care unit, an exspected average of 2 days
  Signals are measured by EEG Monitor and Delir Monitor software
Depth of sedation | At time of surgery and Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
  Intraoperatively: Observe´s Assessment of Alertness/Sedation scale (OAA/S) and postoperatievly: Richmond Agitation Sedation Scale (RASS)
Pain Scales | 3 months
  Perioperatively: Pain sensitivity questionnare; Pain Catastrophing Scale (PCS-GE)(PSQ); Numerische Rating Scale (NRS-V); Behavioural Pain Scale (BPS for ventilated) and BPS-NI (for non-ventilated) patients, Critical-Care Pain Observation Tool (CPOT); Rotterdam Elderly Pain Observation Scale (REPOS); Pupillometry by Neurolight; Intraoperatively: Measurement of the nociceptive flexion reflex threshold (Dolosys Paintracker); Measurement of the pupillary dilation reflex threshold (AlgiScan); Automatic collection of the data of the medication pumps; Multiple blood analysis to measure the plasma-concentrations of anesthetics; Automatic collection of the data of the SED-Line-EEG-Monitor.
Quality indicators of intensive care unit | Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
  Study Center Berlin: This endpoint aims to analyse economic effects of the prospective study patients and retrospective control subjects in the intensive care unit that are caused by the implementation of quality indicators in health care.
Glucosevariability | At time of surgery and Participants will be followed for the duration of intensive care unit stay, an expected average of 5 days
  Measured by Continuous Glucose Monitoring System
Frailty | 3 months, 1, 2 and 5 years after the operation
Coagulationdisorder of the blood | 3 months
  Kidney marker

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charité - University Medicine Berlin; Georg Winterer (BioCog Research Program Coordinator), MD, PhD, Study Chair — Department of Anesthesiology and Intensive Care Medicine, CVK/CCM, Charité - University Medicine Berlin
Locations (2):
- Department of Anesthesiology and Intensive Care Medicine, CCM and CVK, Charité - Universitätsmedizin Berlin, Berlin, Germany
- Department of Intensive Care Medicine, University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Feinkohl I, Hadzidiakos D, Dschietzig TB, Janke J, Heinrich M, Slooter AJC, Spies C, Winterer G, Pischon T. Low-grade, systemic inflammation and the risk of perioperative neurocognitive disorders in an observational study of older adults. Sci Rep. 2025 Dec 20;15(1):44231. doi: 10.1038/s41598-025-31986-z. PMID 41419753
- [Derived] Morgeli R, Borchers F, Feinkohl I, Piper SK, Pischon T, Slooter AJC, Spies C, Wiebach J, Winterer G, Zacharias N, Lammers-Lietz F. A secondary analysis of cortical atrophy and plasma amyloid beta patterns in older patients with cognitive frailty undergoing elective surgery. BMC Geriatr. 2025 Jul 2;25(1):484. doi: 10.1186/s12877-025-05740-z. PMID 40604523
- [Derived] Starks SCE, Pohrt A, Halzl-Yurek F, Heinrich M, Muller A, Spies CD, Winterer G, Zacharias N. Long-term and pre-operative benzodiazepine use in older adults and risk for postoperative delirium: An additional analysis of the multicentre Biomarker Development for Postoperative Cognitive Impairment in the Elderly Study. Eur J Anaesthesiol. 2025 Aug 1;42(8):704-713. doi: 10.1097/EJA.0000000000002201. Epub 2025 May 16. PMID 40384317
- [Derived] Heinrich M, Spies C, Borchers F, Feinkohl I, Pischon T, Slooter AJC, von Haefen C, Zacharias N, Winterer G, Lammers-Lietz F. Perioperative Levels of IL8 and IL18, but not IL6, are Associated with Nucleus Basalis Magnocellularis Atrophy Three Months after Surgery. J Neuroimmune Pharmacol. 2024 Mar 14;19(1):10. doi: 10.1007/s11481-024-10110-4. PMID 38483732
- [Derived] Fislage M, Winzeck S, Woodrow R, Lammers-Lietz F, Stamatakis EA, Correia MM, Preller J, Feinkohl I, Hendrikse J, Pischon T, Spies CD, Slooter AJC, Winterer G, Menon DK, Zacharias N; BioCog Consortium. Structural disconnectivity in postoperative delirium: A perioperative two-center cohort study in older patients. Alzheimers Dement. 2024 Apr;20(4):2861-2872. doi: 10.1002/alz.13749. Epub 2024 Mar 7. PMID 38451782
- [Derived] Trauzeddel RF, Rothe LM, Nordine M, Dehe L, Scholtz K, Spies C, Hadzidiakos D, Winterer G, Borchers F, Kruppa J, Treskatsch S. Influence of a chronic beta-blocker therapy on perioperative opioid consumption - a post hoc secondary analysis. BMC Anesthesiol. 2024 Feb 27;24(1):80. doi: 10.1186/s12871-024-02456-2. PMID 38413849
- [Derived] Fislage M, Feinkohl I, Borchers F, Heinrich M, Pischon T, Veldhuijzen DS, Slooter AJC, Spies CD, Winterer G, Zacharias N; BioCog Consortium. Trail making test B in postoperative delirium: a replication study. BJA Open. 2023 Nov 3;8:100239. doi: 10.1016/j.bjao.2023.100239. eCollection 2023 Dec. PMID 37954892
- [Derived] Fislage M, Feinkohl I, Borchers F, Pischon T, Spies CD, Winterer G, Zacharias N; BioCog Consortium. Preoperative thalamus volume is not associated with preoperative cognitive impairment (preCI) or postoperative cognitive dysfunction (POCD). Sci Rep. 2023 Jul 20;13(1):11732. doi: 10.1038/s41598-023-38673-x. PMID 37474784
- [Derived] Feinkohl I, Janke J, Slooter AJC, Winterer G, Spies C, Pischon T; BioCog Consortium. Metabolic syndrome and the risk of postoperative delirium and postoperative cognitive dysfunction: a multi-centre cohort study. Br J Anaesth. 2023 Aug;131(2):338-347. doi: 10.1016/j.bja.2023.04.031. Epub 2023 Jun 20. PMID 37344340
- [Derived] Ditzel FL, van Montfort SJT, Vernooij LM, Kant IMJ, Aarts E, Spies CD, Hendrikse J, Slooter AJC, van Dellen E; Biomarker Development for Postoperative Cognitive Impairment in the Elderly Consortium. Functional brain network and trail making test changes following major surgery and postoperative delirium: a prospective, multicentre, observational cohort study. Br J Anaesth. 2023 Feb;130(2):e281-e288. doi: 10.1016/j.bja.2022.07.054. Epub 2022 Oct 17. PMID 36261307
- [Derived] Bosancic Z, Spies CD, Muller A, Winterer G, Piper SK, Heinrich M; BioCog Consortium. Association of cholinesterase activities and POD in older adult abdominal surgical patients. BMC Anesthesiol. 2022 Sep 16;22(1):293. doi: 10.1186/s12871-022-01826-y. PMID 36114455
- [Derived] Windmann V, Dreier JP, Major S, Spies C, Lachmann G, Koch S. Increased Direct Current-Electroencephalography Shifts During Induction of Anesthesia in Elderly Patients Developing Postoperative Delirium. Front Aging Neurosci. 2022 Jun 28;14:921139. doi: 10.3389/fnagi.2022.921139. eCollection 2022. PMID 35837483
- [Derived] Fislage M, Feinkohl I, Pischon T, Spies CD, Borchers F, Winterer G, Zacharias N; BioCog Consortium. Presurgical Thalamus Volume in Postoperative Delirium: A Longitudinal Observational Cohort Study in Older Patients. Anesth Analg. 2022 Jul 1;135(1):136-142. doi: 10.1213/ANE.0000000000005987. Epub 2022 Jun 16. PMID 35442218
- [Derived] Lammers-Lietz F, Zacharias N, Morgeli R, Spies CD, Winterer G. Functional Connectivity of the Supplementary and Presupplementary Motor Areas in Postoperative Transition Between Stages of Frailty. J Gerontol A Biol Sci Med Sci. 2022 Dec 29;77(12):2464-2473. doi: 10.1093/gerona/glac012. PMID 35040961
- [Derived] Heinrich M, Sieg M, Kruppa J, Nurnberg P, Schreier PH, Heilmann-Heimbach S, Hoffmann P, Nothen MM, Janke J, Pischon T, Slooter AJC, Winterer G, Spies CD. Association between genetic variants of the cholinergic system and postoperative delirium and cognitive dysfunction in elderly patients. BMC Med Genomics. 2021 Oct 21;14(1):248. doi: 10.1186/s12920-021-01071-1. PMID 34674705
- [Derived] Koch S, Windmann V, Chakravarty S, Kruppa J, Yurek F, Brown EN, Winterer G, Spies C; BioCog Study Group. Perioperative Electroencephalogram Spectral Dynamics Related to Postoperative Delirium in Older Patients. Anesth Analg. 2021 Dec 1;133(6):1598-1607. doi: 10.1213/ANE.0000000000005668. PMID 34591807
- [Derived] Lichtner G, Zacharias N, Spies CD, Feinkohl I, Winterer G, Pischon T, von Dincklage F; BioCog Consortium. Resting state brain network functional connectivity is not associated with inflammatory markers and blood cell counts in older adults. Clin Neurophysiol. 2021 Jul;132(7):1677-1686. doi: 10.1016/j.clinph.2021.03.042. Epub 2021 May 2. PMID 34044190
- [Derived] Heinrich M, Muller A, Cvijan A, Morgeli R, Kruppa J, Winterer G, Slooter AJC, Spies CD; BioCog Consortium. Preoperative Comparison of Three Anticholinergic Drug Scales in Older Adult Patients and Development of Postoperative Delirium: A Prospective Observational Study. Drugs Aging. 2021 Apr;38(4):347-354. doi: 10.1007/s40266-021-00839-5. Epub 2021 Mar 15. PMID 33721289
- [Derived] Kant IMJ, de Bresser J, van Montfort SJT, Mutsaerts HJMM, Witkamp TD, Buijsrogge M, Spies C, Hendrikse J, Slooter AJC. Preoperative brain MRI features and occurrence of postoperative delirium. J Psychosom Res. 2021 Jan;140:110301. doi: 10.1016/j.jpsychores.2020.110301. Epub 2020 Nov 16. PMID 33260072
- [Derived] Deffland M, Spies C, Weiss B, Keller N, Jenny M, Kruppa J, Balzer F. Effects of pain, sedation and delirium monitoring on clinical and economic outcome: A retrospective study. PLoS One. 2020 Sep 2;15(9):e0234801. doi: 10.1371/journal.pone.0234801. eCollection 2020. PMID 32877411
- [Derived] van Montfort SJT, van Dellen E, Wattel LL, Kant IMJ, Numan T, Stam CJ, Slooter AJC. Predisposition for delirium and EEG characteristics. Clin Neurophysiol. 2020 May;131(5):1051-1058. doi: 10.1016/j.clinph.2020.01.023. Epub 2020 Feb 21. PMID 32199395
- [Derived] Feinkohl I, Borchers F, Burkhardt S, Krampe H, Kraft A, Speidel S, Kant IMJ, van Montfort SJT, Aarts E, Kruppa J, Slooter A, Winterer G, Pischon T, Spies C. Stability of neuropsychological test performance in older adults serving as normative controls for a study on postoperative cognitive dysfunction. BMC Res Notes. 2020 Feb 4;13(1):55. doi: 10.1186/s13104-020-4919-3. PMID 32019577
- [Derived] Kant IMJ, Mutsaerts HJMM, van Montfort SJT, Jaarsma-Coes MG, Witkamp TD, Winterer G, Spies CD, Hendrikse J, Slooter AJC, de Bresser J; BioCog Consortium. The association between frailty and MRI features of cerebral small vessel disease. Sci Rep. 2019 Aug 5;9(1):11343. doi: 10.1038/s41598-019-47731-2. PMID 31383903
- [Derived] Windmann V, Spies C, Brown EN, Kishnan D, Lichtner G, Koch S; BioCog Study Group. Influence of midazolam premedication on intraoperative EEG signatures in elderly patients. Clin Neurophysiol. 2019 Sep;130(9):1673-1681. doi: 10.1016/j.clinph.2019.05.035. Epub 2019 Jul 10. PMID 31351371
- [Derived] Lachmann G, Kant I, Lammers F, Windmann V, Spies C, Speidel S, Borchers F, Hadzidiakos D, Hendrikse J, Winterer G, de Bresser J; BIOCOG Consortium. Cerebral microbleeds are not associated with postoperative delirium and postoperative cognitive dysfunction in older individuals. PLoS One. 2019 Jun 14;14(6):e0218411. doi: 10.1371/journal.pone.0218411. eCollection 2019. PMID 31199858
- [Derived] Feinkohl I, Janke J, Hadzidiakos D, Slooter A, Winterer G, Spies C, Pischon T. Associations of the metabolic syndrome and its components with cognitive impairment in older adults. BMC Geriatr. 2019 Mar 7;19(1):77. doi: 10.1186/s12877-019-1073-7. PMID 30845934